CLINICAL TRIAL: NCT01365117
Title: Phase 1, Single-center, Open-label, Randomized, Crossover Design Clinical Trial in Healthy Normal Volunteers to Evaluate Insulin Exposure and Dose-proportionality Following Inhalation of Technosphere® Insulin Inhalation Powder (3 U and 4 U Insulin/mg) Using the Gen2 Inhaler
Brief Title: Pharmacokinetic Study in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-167
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2012-06-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: Technosphere® Insulin Inhalation Powder
- Cohort 2 (Experimental)
  Interventions: Drug: Technosphere® Insulin Inhalation Powder

INTERVENTIONS:
Drug: Technosphere® Insulin Inhalation Powder — 15 subjects in a three-way crossover (three different doses of TI Inhalation Powder [one 20 U, two 20 U and one 40 U cartridges)
  Other Names: Inhaled human insulin and Technosphere Powder
  Arms: Cohort 1
Drug: Technosphere® Insulin Inhalation Powder — 16 subjects in a four-way crossover (four different doses of TI Inhalation Powder [one 20 U, one 20 U plus one 10U, one 30 U (3 U per mg), one 30 U (4 U per mg cartridges)])
  Other Names: Inhaled human insulin and Technosphere Powder
  Arms: Cohort 2

SUMMARY:
Phase 1 clinical trial to evaluate insulin exposure using different formulations of Technosphere Insulin Inhalation Powder using the Gen2 inhaler in healthy normal volunteers.

DETAILED DESCRIPTION:
Phase 1, single-center, open-label, randomized, crossover clinical trial to evaluate insulin exposure using the 3 U/mg and 4 U/mg Technosphere Insulin Inhalation Powder formulations administered using the Gen2 inhaler in 31 healthy volunteers. Drop outs will be replaced. Each subject will undergo a screening visit and either 4 or 5 days of in clinic stay and dosing, depending on randomization schedule.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking (within the last 6 months) men and women aged 18 to 45 years who are considered healthy
* Body mass index (BMI) < 32 kg/m2
* FEV1 ≥ 80% of the Third National Health and Nutrition Examination Survey (NHANES III) predicted

Exclusion Criteria:

* Pre-existing asthma or chronic obstructive pulmonary disease (COPD)
* History of coronary artery disease, peripheral vascular disease, or congestive heart failure
* Blood donation within the previous 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2011-01; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The relative exposure (Cmax and AUC0-120) of insulin from TI Inhalation Powder as delivered | 0-120 minutes

SECONDARY OUTCOMES:
Safety will be assessed by adverse events | 32 days
Safety will be assessed by Spirometry (FEV1) | 32 Days
Safety will be assessed by vital sign measurements | 32 Days
Safety will be assessed by physical examination findings. | 32 Days
Safety will be assessed by clinical laboratory test results. | 32 Days

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Connolly, M.D., Principal Investigator — Celerion
Locations (1):
- Celerion, Neptune City, New Jersey, United States